CLINICAL TRIAL: NCT05187429
Title: Safety, Immunogenicity and Efficacy of Low Dose Nivolumab in Adults Living With HIV on Antiretroviral Therapy (ART)
Brief Title: Low Dose Nivolumab in Adults Living With HIV on Antiretroviral Therapy
Acronym: NIVO-LD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: The Alfred (Other); NCID (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 358/20
Record Dates: First submitted 2021-12-15; First posted 2022-01-11 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: HIV I Infection
Keywords: HIV; Antiretroviral interruption; ATI; Low dose Nivolumab; Clinical Trial
MeSH Terms: interventions — Nivolumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: In Part 1 (Cohort A) - there is no masking and the Nivolumab administered is open-labeled. There is no randomization in this group.
  In Part 2 (Cohort B) - the participant, care provider and investigator are all masked to the treatment allocation. Participants in this group will be assigned to intervention treatment by chance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose escalation phase (Cohort A) (Experimental): Drug: Nivolumab Dose form: infusion Dose route: intravenous Dosage: 0.1, 0.3 or 1.0 mg/kg Duration: Single dose administered on Study Day 7
  Interventions: Drug: Nivolumab 10 MG/ML [Opdivo]
- Randomization phase (Cohort B) (Experimental): Drug: Nivolumab Dose form: infusion Dose route: intravenous Dosage: 1.0mg/kg (determined from Cohort A) Duration: single dose administered on Day 0 (baseline)
  Interventions: Drug: Nivolumab 10 MG/ML [Opdivo]
- Randomization phase comparator (Cohort B) (Placebo Comparator): Drug: Nivolumab Comparator: saline Dose form: infusion Dose route: intravenous Dosage: 1.0mg/kg of Nivolumab Duration: single dose administered on Day 0 (baseline)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Nivolumab 10 MG/ML [Opdivo] — Cohort A: Dose escalation phase: Nivolumab will be administered intravenously as a single dose in the dose escalation phase.
  Arms: Dose escalation phase (Cohort A)
Drug: Nivolumab 10 MG/ML [Opdivo] — Cohort B: Randomization phase: Nivolumab will be administered intravenously as a fixed single dose (1.0 mg/kg) in the randomization phase.
  Arms: Randomization phase (Cohort B)
Drug: Saline — Cohort B: Randomisation phase: Saline will be administered intravenously as a single dose in the randomisation arm.
  Arms: Randomization phase comparator (Cohort B)

SUMMARY:
The purpose of this study is to evaluate whether a single dose of Nivolumab in people living with HIV can reduce the latent reservoir. The latent HIV reservoir is a group of immune system cells in the body that are infected with HIV but are not actively producing new virus. This is the reason why people living with HIV are unable to stop their antiretroviral treatment.

DETAILED DESCRIPTION:
This study consists of 2 Parts.

Part 1 is a dose escalation phase. This phase is open-label, single dose titration study in adult people living with HIV. There are 3 stages: a screening stage of up to 14 days; on study study treatment stage, where Nivolumab will be administered on Day 7 and a follow-up stage of up to 168 days (6 months), depending on the dose level. The maximum total duration on study for each participant enrolled in this phase is 140 days (6.3 months).

Part 2 is a double-blind, randomized, placebo controlled clinical trial of a single fixed dose of 1.0mg/kg Nivolumab administered intravenous (IV) infusion compared with placebo in adult people living with HIV. This part of the study will consist of 3 stages: a screening stage of up to 21 days; on study study treatment stage, where Nivolumab/placebo will be administered on Day 0, followed by a maximum of 6months of an analytical treatment interruption (where antiretroviral therapy (ART) is ceased), before the participant re-commences ART. The maximum total duration on study for each participant enrolled in this phase is 241 days (approximately 8 months).

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection;
* Viral load > 400 copies/mL prior to initiation of ART;
* Weight ≥ 50 kg;
* Ability and willingness to provide informed consent and to continue ART throughout the study;
* Receiving combination ART for at least 2 years and being on the same ART regimen for at least 4 weeks at the screening visit;
* HIV-1 plasma RNA <50 copies/mL for >2 years (documented on at least 2 occasions within the 2 years) and <50 copies/mL at screening. Episodes of a single HIV plasma RNA 50-500 copies/mL will not exclude participation if the subsequent HIV plasma RNA was <50 copies/mL;
* CD4+ T cell counts >500 cells/μL at screening;
* Female participants if they meet one of the following criteria:

  * Is of non-child-bearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or,
  * Is of child-bearing potential with a negative pregnancy test at both Screening and Day 0 and agrees to use one of the following methods of contraception to avoid pregnancy from 14 days prior to the first infusion until the end of the study:

    * Complete abstinence from penile-vaginal intercourse;
    * Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide);
    * Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year;
    * Male partner sterilization confirmed prior to the female participant's entry into the study, and this male is the sole partner for that participant;
    * Approved hormonal contraception (Where other medications to be used in the study (e.g., efavirenz and darunavir) are known, or are likely, to significantly interact with systemic contraceptives, resulting in decreased efficacy of the contraceptive, then alternative methods of non-hormonal contraception are recommended);
    * Any other method with published data showing that the expected failure rate is <1% per year. Note: If using one of the described contraception methods it must be used consistently, in accordance with the approved product label and all female participants must be willing to undergo urine pregnancy tests as specified in the Schedule of Procedures.
* All participants must agree not to participate in a conception process (e.g. active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization, egg donation) during the study;
* Heterosexually active male if they are;

  * willing to use an effective method of contraception (anatomical sterility in self that is confirmed prior to study entry) or
  * agree on the use of an effective method of contraception with an effective failure rate of < 1% by his partner (hormonal contraception, intra-uterine device (IUD), or anatomical sterility) from the day of the first infusion until the end of study (as long as plasma viral load <20c/mL).
* Singapore only: all participants must understand and agree to abide by the Infectious Diseases Act, in particular Part 4 'Control of HIV infection' inclusive of section 23 'Sexual activity by person with HIV infection'

Exclusion Criteria:

* Active, known and suspected autoimmune disease (including but not limited to including but not limited to inflammatory bowel diseases, scleroderma, severe psoriasis, myocarditis, uveitis, pneumonitis, systemic lupus erythematosus, rheumatoid arthritis, optic neuritis, myasthenia gravis, adrenal insufficiency, hypothyroidism and/or hyperthyroidism, autoimmune thyroiditis, sarcoidosis, and vitiligo);
* History of interstitial lung disease;
* History of chronic obstructive pulmonary disease (COPD);
* Type I diabetes mellitus;
* Active malignancy or history of malignancy requiring systemic chemotherapy or surgery in the preceding 24 months; exception -history of excised localized non-melanomatous skin cancers (squamous cell carcinoma, basal cell carcinoma);
* History of solid organ transplant. Note Individuals with prior corneal transplants may be allowed to enroll after discussion with and approval from the study principal investigator;
* Active or previously treated active TB;
* History of HIV-related opportunistic infection within the last years prior to study entry;
* Prior history of immune reconstitution syndrome (IRIS);
* Current, chronic, acute or recurrent bacterial, fungal or viral (other than HIV) infections that are serious, in the opinion of the investigator, and require systemic therapy within 30 days prior to study entry;
* Immune deficiency other than that caused by HIV infection;
* Received investigational drug or device within 6 months prior to study entry
* Treatment for hepatitis C virus (HCV) within 6 months prior to study entry;
* History of previous treatment with an immune checkpoint inhibitor;
* History of prior immunoglobulin (IgG) therapy;
* Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), systemic cytotoxic chemotherapy, experimental vaccines or investigational therapy within 60 days prior to study entry or intent to use immunomodulators during the study. NOTE: Participants receiving stable physiologic glucocorticoid doses, defined as prednisolone less than or equal to 10 mg/day or the equivalent, will not be excluded. Stable physiologic glucocorticoid doses should not be discontinued for the duration of the study. In addition, participants receiving inhaled or topical corticosteroids will not be excluded;
* Any other current or prior therapy which, in the opinion of the investigators, would make the individual unsuitable for the study or influence the results of the study;
* Participants with severe hepatic impairment (Class C) as determined by Child-Pugh classification;
* Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones);
* Participants who intend to modify their ART regimen within the study period;
* Active alcohol or substance use that in the opinion of the investigator will prevent adequate compliance with study procedures;
* Any acute or chronic psychiatric problems that, in the opinion of the investigator, make the participant ineligible for participation;
* Any active, clinically significant medical condition not otherwise covered;
* Women who are pregnant or breastfeeding or Women of Child Bearing Potential (WOCBP) who are unwilling or unable to use an acceptable method of contraception to avoid pregnancy as specified in the inclusion criteria;
* Men of reproductive potential who are unwilling or unable to use an acceptable method of contraception to avoid pregnancy as specified in the inclusion criteria;
* Specific exclusion criteria for Cohort A (Fine Needle Biopsy):

  * prothrombin time (PTT) >2x ULN
  * international normalized ratio (INR) >1.5
  * Platelets <50,000/mm3
  * Chronic venous stasis of lower extremities
  * Lower extremity lymphedema
  * Allergies to local anesthetic
  * Blood coagulation disorder.
* The following laboratory abnormalities (lab tests may be repeated to obtain acceptable values before failure at screening is concluded);

  * Hematology:

    * Hemoglobin < 14.0 g/dL for men and <12.0 g/dL for women;
    * Absolute Neutrophil Count (ANC) ≤ 1,500 /mm^3 (≤ 1 x 10^9/L);
    * Platelets ≤ 150,000 /mm^3
  * Biochemistry:

    * Aspartate aminotransferase (AST) > 1.25 x ULN;
    * Alanine aminotransferase (ALT) > 1.25 x ULN;
    * Bilirubin ≥1.5 x ULN (if on atazanavir ≥5 x ULN);
    * Interferon-gamma release assay (IGRA) for tuberculosis (TB) with negative results within 90 days prior to study entry
    * Thyroid stimulating hormone (TSH) outside the normal reference range;
    * Free thyroxine (T4) outside the normal reference range
    * Presence of Anti-thyroid peroxidase (TPO) antibodies;
    * Presence of anti-glutamic acid decarboxylase (GAD) antibodies
    * Antinuclear antibody (ANA) >1:80 at screening
    * Early morning (8-9 am) cortisol outside the normal reference range. Note: female participants on estrogen-containing oral contraception or other exogenous estrogen treatment may repeat the AM cortisol as part of screening to determine eligibility;
    * Fasting blood sugar > 7.0 mmol/L (unless already diagnosed with Type 2 Diabetes Mellitus);
  * Microbiology:

    * Positive for hepatitis B surface antigen;
    * Positive for hepatitis C antibody, unless confirmed clearance of HCV infection (spontaneous or following treatment) by polymerase chain reaction (PCR) testing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events enrolled in Cohort A | 23 weeks
  Incidence and severity of Adverse Events (defined as Common Terminology Criteria (CTC) grade 3 or higher according to the Division of AIDS (DAIDS) grading table) that are definitely, probably or possibly related to study treatment during the study period
Number of participants with treatment-emergent adverse events enrolled in Cohort B | 31 weeks
  Incidence and severity of Adverse Events (defined as CTC grade 3 or higher according to the DAIDS grading table) that are definitely, probably or possibly related to study treatment during the study period

SECONDARY OUTCOMES:
Change in PD-1 receptor occupancy in peripheral blood following a single low dose of nivolumab in participants enrolled in Cohort A | Day 7, Day 14, Day 21, Day 35, Day 63, Day 91, Day 126, Day 168
  Time course change in the percentage PD-1 receptor occupancy on T-cells in peripheral blood determined by flow cytometry. Nivolumab infusion occurs on Day 7 study visit. Day 168 timepoint only applicable to 1.0mg/kg cohort
Change in PD-1 receptor occupancy in lymph node T-cells following a single low dose of nivolumab in participants enrolled in Cohort A. | Day 0, Day 21
  Time course change in the percentage PD-1 receptor occupancy on T-cells in inguinal lymph node T-cells determined by flow cytometry
Cohort A: T-cell responses to Gag peptides | Day 0, Day 126
  Number of cluster of differentiation 4 (CD4) and/or cluster of differentiation 8 (CD8) T-cells responses to Gag peptides by intracellular cytokine staining both in peripheral blood and lymph nodes
Cohort A: T-cell responses to Pol/Env/Nef peptides | Day 0, Day 126
  Number of CD4 and/or CD8 T-cells responses to Pol/Env/Nef peptides by intracellular cytokine staining in both peripheral blood and lymph nodes
Change in PD-1 receptor occupancy in peripheral blood following a single low dose of nivolumab in participants enrolled in Cohort B | Day 0, Day 7, Day 28, Day 168
  Time course change in the percentage PD-1 receptor occupancy on T-cells in peripheral blood determined by flow cytometry. Nivolumab/placebo infusion occurs on Day 0 (baseline) visit
Cohort B: HIV RNA | 24 weeks
  Proportion of participants with a viral load (HIV RNA) > 50 and > 1000c/ml measured weekly during an ART interruption, which starts on Day 7 and ends at a maximum of week 24 (earlier if ART re-start criteria are met)
Cohort B: viral rebound | 24 weeks
  Number of participants who experience a viral rebound (defined as first viral load > 50 copies/mL) during an ATI period which starts on Day 7 and ends at a maximum of week 24 (earlier if ART re-start criteria are met).
Cohort B: T-cell responses to Gag peptides | Day 7, Day 168
  Number of CD4 and/or CD8 T-cells responses to Gag peptides by intracellular cytokine staining both in peripheral blood and lymph nodes
Cohort B: T-cell responses to Pol/Env/Nef peptides | Day 7, Day 168
  Number of CD4 and/or CD8 T-cells responses to Pol/Env/Nef peptides by intracellular cytokine staining in both peripheral blood and lymph nodes

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Lewin, Principal Investigator — University of Melbourne
Locations (2):
- Alfred Hospital - Department of Infecious Diseases, Melbourne, Victoria, Australia
- Tan Tock Seng Hospital, Singapore, Singapore